CLINICAL TRIAL: NCT07353255
Title: Flexible Fibrescope Versus Video Laryngoscope for Nasotracheal Intubation - A Randomised Comparison
Brief Title: Fibrescope vs Videolaryngoscope for Nasotracheal Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 343162
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: No Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Fibrescope (Active Comparator): Randomly allocated to have intubation using flexible fibrescope
  Interventions: Device: Nasotracheal Intubation with Fibrescope
- Videolarygoscope (Active Comparator): randomly allocated to have intubation using videolaryngocope
  Interventions: Procedure: Nasotracheal Intubation with Video laryngoscope

INTERVENTIONS:
Device: Nasotracheal Intubation with Fibrescope — Intubation of trachea via nasal route with Fibrescope (11302BDX Flex. Intubation Video Endoscope 4 x 65 Karl Storz)
  Arms: Flexible Fibrescope
Procedure: Nasotracheal Intubation with Video laryngoscope — Intubation of trachea via nasal route using a videolaryngoscope (301-000-000 McGRATH™ with Mac Blade)
  Arms: Videolarygoscope

SUMMARY:
Patients having surgery under general anaesthesia require insertion of a breathing tube to keep the airway open. The technique of inserting a breathing tube through the nose into the trachea (airway) is known as nasotracheal intubation. This is the ideal airway for surgical procedures performed inside the mouth such as complex teeth extractions and operations on the jaw.

Traditionally, the breathing tube is initially inserted blindly into the nasal cavity, then a video laryngoscope (a camera device) or a direct laryngoscope is used to visualise and guide the passage of tube into the trachea. This approach can be associated with difficulty passing the tube and a has high incidence of nasal trauma and nosebleed. A flexible fibrescope ( flexible camera device) with pre-loaded tracheal tube is passed through the nostril first under vision, gently advanced through the nasal passage and then to the trachea. Once it is correctly placed in the trachea, the breathing tube is railroaded over it. This procedure allows to visualise the nasal passage and to choose most patent nostril and hence likely to reduce risk of nosebleed as compared blind passage of tube through the nose. A videolaryngoscope has a camera on the blade that projects the image onto a monitor screen. As this is a rigid device, it can only be inserted through the oral cavity and allows the advancement of tube into the trachea. Both these techniques are currently used in the clinical practice. However, there are no studies to inform the anaesthetists whether there are any differences in the incidence of nosebleed.

We wish to do a randomised comparison between flexible fibrescope and videolaryngocope in terms reducing the risk and severity of nosebleed.

Patients aged 18 and above, presenting for elective surgical procedures and requiring general anaesthesia and nasal intubation will be invited to take part in the study. We are aiming to recruit 200 participants (see sample size section) to see any significant differences in the incidence of nosebleed.

Patients who are eligible and consent to take part in the study will be randomly allocated either to flexible fibrescope group or to videolaryngoscope. At the time of nasotracheal intubation, smoothness of nasal intubation, severity of bleeding from the nose and time taken to complete the tracheal intubation will be noted. Five minutes after intubation, the surgeon performing surgery (blinded to the technique of intubation) will be examining the oral cavity for any bleeding. This will be graded using a standardised nasal bleeding score. All patients will be visited in the post operative period to check any ongoing nosebleed and nasal discomfort. Patient details that will be collected includes gender, age, weight, height, body mass index and airway assessment parameters. No other personal data is required.

This study aims to see whether the use of flexible fibrescope reduces nasal bleeding and improves patient safety. If there is no difference, it may provide reassurance in the continued use of video laryngoscopy for nasal intubation.

DETAILED DESCRIPTION:
STUDY PROTOCOL

FLEXIBLE FIBRESCOPE VERSUS VIDEOLARYNGOSCOPE FOR NASOTRACHEAL INTUBATION- A RANDOMISED COMPARISON

1. INTRODUCTION The technique of inserting a tracheal tube through the nasal passage into the trachea (airway) is known as nasotracheal intubation. This is the preferred airway for surgical procedures performed in and around oral cavity including dental procedures. Traditionally, the tracheal tube is initially inserted blindly into the nasal cavity. A laryngoscope is then used to visualise and help guide the passage of the tube into the trachea. This approach can be associated with difficulty passing the tube and a high incidence of nasal trauma [1, 2], as the nasal passages can be narrow and demonstrate inter-individual anatomic variability. Therefore, various approaches have been described in the literature to reduce nasal trauma including warming the tube [3], applying water-based lubricants and preparing the nasopharynx with progressive dilation and/or a topical vasoconstrictors [4]. There have been randomised studies using curve-tipped suction catheters [2], and bougies [1,5] showing reduced incidence of nasal trauma as compared to blind passage of the tube through the nose. However, as these devices are blindly inserted through the nasal passage, the device itself can cause some degree of trauma. Using a fiberscope allows for an assessment of the patency of the nasal passages and visualisation of the path the tube will take through the nasopharynx. We therefore hypothesise that using a flexible fiberscope for nasal intubation will reduce nasal trauma.

   A flexible fiberscope (A in Figure below) is a device that employs flexible fibreoptic bundles to allow the transmission of an image via internal reflection of light. The image is then transmitted to an external screen. These devices were first used in the 1950's and allow successful intubation of the trachea for both anticipated and unanticipated difficult airways [6].

   A video laryngoscope has a camera on the blade that projects the image onto a monitor screen (B in Figure below). This means that the person intubating can see around the corner and get a better view of the vocal cords. Unlike a flexible fiberscope, video laryngoscopes can only be inserted through the mouth and therefore can't visualise the nasal passages. Therefore, passage of the tube through the nasal passage is blind when video laryngoscopy is used for nasal intubation.

   1.1 Background For surgical procedures in and around the oral cavity (dental and maxillo-facial surgery), tracheal intubation via the nasal route allows optimal access and facilitates surgery. Use of bougies and catheters have been described in the literature to improve success rates and reduce nasal tissue trauma during nasotracheal intubation [1, 2, 5]. However, in these studies devices such as catheters or bougies, were inserted blindly through the nasal passage. Use of a flexible fibrescope eliminates blind insertion of any device via nasal passage and in addition, allows assessment to inform an objective choice of the best nasal passage (right vs left) to use for intubation.

   1.2 Proposed study We hypothesise that the use of the flexible fibrescope will reduce the incidence of nasal trauma when compared to a video laryngoscope.

   1.3 Study population Patients aged above 18, presenting for elective surgical procedures and requiring nasotracheal intubation will be invited to take part in the study.

   1.4 Treatment/Intervention On arrival to theatre, following a standard WHO surgical safety check list, patients will be randomly allocated to either flexible fibrescope or video laryngoscope to facilitate nasotracheal intubation. All patients will receive decongestant nasal spray of 5% lidocaine with 0.5% phenylephrine 1 ml in each nostril. The rest of the anaesthetic management will remain normal as planned by the lead anaesthetist. During nasotracheal intubation the data collected will include severity of nasal trauma on a 4 point scale (Appendix 1), smoothness of nasal intubation on a 4 point scale (Appendix 1), laryngoscopy time (from insertion of laryngoscope in the mouth to visualize the vocal cords or from insertion of fiberscope in the nostril to visualise the vocal cords), intubation time (time from insertion of fiberscope or video laryngoscope till first capnography trace) and first attempt success rate (% of intubations succeeded in first attempt), number of intubation attempts and any additional manoeuvres required (external pressure on thyroid cartilage, tube rotation, tube impingement).

   1.5 Pre-clinical data In three studies [1,2, 3, 5], time to nasal intubation and severity of nasal trauma were all reduced by utilising either a bougie or suction catheter with or without a nasopharyngeal airway.

   1.6 Clinical Data Both flexible fibrescopes and video laryngoscopes are routinely used in clinical practice at University Hospitals Coventry and Warwickshire NHS Trust for nasotracheal intubation.
2. RATIONALE 2.1 Aims and hypothesis We hypothesise that the use of the flexible fibrescope will reduce nasal trauma and bleeding whilst improving first time intubation success rates when compared to video laryngoscope-assisted nasal intubation.

   2.2 Justification

   Trauma during nasotracheal intubation is commonly described in the literature and can range from minor epistaxis to significant damage and dissection of the nasal cavity and secondary bacteraemia [1,2, 3, 5,]. This can occur because the nasal cavity is highly vascular and contains space limiting folds named 'turbinates' and 'conchae', that play an important physiological role in warming and humidifying air, which can also become obstructed due to infections and or allergies. The nasal cavity also often contains abnormalities and variations such as septal deviation, polyps, concha bullosa, septal spurs, stenosis, and choanal atresia [8]. Passage of a tube through the nasal cavity can therefore easily lead to nasal trauma and reduce success rate of nasal intubation. Various approaches have therefore been described in the literature to reduce nasal trauma. Techniques such as warming the tube [3], applying water-based lubricants, preparing the nasopharynx with progressive dilation and/or a topical vasoconstrictor [4] have been applied with varying success. Use of curve-tipped suction catheters [2], and bougies [1,5] as a guide to nasal tubes have been shown to reduce nasal trauma.

   In current practice both flexible fibrescopes and video laryngoscopes are routinely used for tracheal intubation. However, with video laryngoscopy during nasal intubation, insertion of tube through the nasal passage is blind. Therefore, some practitioners prefer using a fiberscope for nasal intubation. Clinicians are uncertain as to which is the best approach. To our knowledge, previous studies have not utilised flexible fibrescopes to eliminate blind insertion of the tube in the nostril. Comparing the efficacy of a flexible fibrescope with a tracheal tube railroaded over it to a video laryngoscope for nasotracheal intubation could inform airway practitioners on their choice of technique to improve success and minimise bleeding risk.

   2.3 Assessment and management of risk For this study, patients requiring general anaesthesia and nasotracheal intubation for elective surgical procedures will be recruited. The flexible fibrescope and video laryngoscope selected for this study are currently used in routine clinical practice as intubation aids. In the event of any unanticipated difficulty with intubation, the lead anaesthetist will follow the Difficult Airway Society guidelines and data collection will stop at this point.

   The lead anaesthetist is free to choose different airway equipment to those specified by the study if they feel that this would be clinically appropriate. We do not anticipate any additional risks to the study participants. During the procedure of airway management, all patients will be closely monitored as specified by 'Association of Anaesthetists' standards of monitoring during anaesthesia. This includes peripheral oxygen saturation, end tidal oxygen, depth of anaesthesia and end-tidal CO2, ECG and blood pressure.
3. OBJECTIVES AND OUTCOME MEASURES/ENDPOINTS

3.1 Primary objective The aim of the study will be to see which of two airway devices (flexible fibrescope or video laryngoscope) is best suited for reducing trauma during nasotracheal intubation.

3.2 Secondary objectives The secondary objectives are to compare factors relating to speed and ease of nasotracheal intubation, along with postoperative patient-centred outcomes such as presence of any sore throat or bleeding between the two groups.

3.3 Primary endpoint/outcome The primary outcome will be incidence and severity of nasal trauma scored using the 'nasal trauma score' 5 minutes post intubation (Appendix 1).

3.4 Secondary endpoints/outcomes

1. Nasal intubation smoothness score (Appendix 1)
2. Total Intubation time
3. Laryngoscopy time
4. Incidence of post operative sore throat
5. Incidence of postoperative nasal discomfort

4. STUDY DESIGN Randomised Controlled trial

On arrival to theatre, following a standard WHO surgical safety check list, patients will be randomly allocated to have nasotracheal intubation either using flexible fiberscope or video laryngoscope.

5. STUDY SETTING This will be a single centre study, conducted at University Hospitals Coventry & Warwickshire NHS Trust

6. ELIGIBILITY CRITERIA Patients scheduled to undergo elective surgical procedures will be assessed for eligibility.

6.1 Inclusion criteria Patients aged 18 and above, presenting for elective surgical procedures and requiring general anaesthesia and nasal intubation will be invited to take part in the study.

6.2 Exclusion criteria · Patients who do not want to take part or do not give consent

· Patients unable to give written consent.

· Patient physical status of ASA 4 and 5,

· Patients deemed to require awake intubation.

7. TRIAL PROCEDURES

Suitable patients for the study will be approached in the preoperative assessment clinic during a face-to-face visit. An invitation letter and patient information sheet will be provided during preoperative assessment. Adequate time will be given to read the patient information sheet. One of the research team members will approach the patient on the day of surgery and answer any queries. If they are satisfied and willing to take part in the study, written consent will be obtained on the day of surgery.

7.1 Recruitment

The chief investigator and co-investigators will identify suitable operating lists based on the scheduled surgical procedures. Only those patients meeting the inclusion criteria will be approached.

7.2 Patient identification

Patients undergoing surgery that requires nasotracheal intubation are suitable for inclusion in the study. Scheduled operating lists will be screened by the chief investigator and principal investigator and suitable patients identified.

During the preoperative assessment, one of the research team members will provide a patient information sheet. Patients will be given adequate time to read the information and any questions will be answered. If they are satisfied and willing to take part in the study, written consent will be obtained on the day of surgery.

7.3 Payment

There is no payment for any participant for taking part in the study

7.4 Consent

Participants will be given adequate time to read and understand the patient information leaflet. Once they have read the information, any questions will be answered. If they agree for the study, they will be asked to complete the consent form. The consent will be obtained by chief investigator, principal investigator or one of the research team members delegated and supervised by the investigators.

7.5 Randomisation scheme

Sample size: Sample size is based on the primary outcome of incidence of nasal bleeding. A previous study of video laryngoscope assisted nasotracheal intubation reported a rate of bleeding detected in the posterior pharynx of 68% (Abrons 2017). A relative reduction in 33% is considered clinically significant. To detect this treatment difference at a significant level of 5% and power of 90%, a total sample of 186 patients is required. To account for failure and loss of follow up, we will recruit a total of 200 patients.

Randomisation Methodology: Participants will be randomised using a paper randomisation list that will be provided to the UHCW Research and Development (R&D) department, independent from the rest of the study team. The randomisation list will be generated by the study statistician prior to recruitment starting. The method of permuted random blocks will be utilised, with varying block sizes used. Sealed opaque randomisation envelops will be stored in a locked research cabinet in the R&D Department. They will be signed out as and when needed.

On arrival in the anaesthetic room, patients will be monitored using peripheral oxygen saturation, end-tidal CO2, depth of anaesthesia, ECG and blood pressure. Patients will be randomly allocated to one of two groups as described below by opening the sealed envelope.

1. Fibrescope group
2. Video laryngoscope group

Both a flexible fiberscope and a video laryngoscope will be available in the anaesthetic room prior to revelation of the group. Once nasotracheal intubation is completed, the rest of the anaesthetic management will proceed as planned by the lead anaesthetist.

All other aspects of patient care outside of the randomisation to fibrescope or video laryngoscopy for nasotracheal intubation will be conducted in accordance with routine clinical practice and local guidelines.

For patients randomised to the video laryngoscope, laryngoscopy will be performed using the video laryngoscope: Mcgrath ™ MAC video laryngoscope (Medtronic Plc, Galway Ireland). A lubricated 6.0 mm ID tube: Polar™ Preformed Tracheal tube, North Nasal Profile™ (Smiths Medical ASD, Inc, Minneapolis, USA) will be inserted through the most patent nostril (as identified during preoperative visit) and advanced until it reaches the posterior nares. It will be then advanced through the vocal cords into the trachea under video guidance. If there was any hold-up immediately after passing the tube through the nostrils, the tube will be gently rotated to allow passage through the nasopharynx. If there is any impingement at the level of arytenoids, the tube will be withdrawn slightly, rotated anticlockwise and then advanced.

For patients randomised to the fiberscope, the same tube type will be loaded on the 4mm fibrescope: Flex. Intubation Video Endoscope 4 x 65 - model 11302BDX (Karl Stortz Tuttlingen, Germany) prior to beginning intubation. The fibrescope will then be inserted into the most patent nostril. If this nostril is deemed to be adequate by the operator, the procedure will continue, otherwise the other nostril will be assessed and the most optimal nostril will be chosen for intubation. The fibrescope will be advanced through the nasopharynx and into the trachea. At this point the tube will be advanced over the fiberscope from the trachea.

Correct placement of the tube will be confirmed using end tidal CO2 and the rest of the anaesthetic management will proceed as planned by the lead anaesthetist. Patients will be followed up from 3 - 24 hours post op to assess for nasal discomfort, sore throat and bleeding.

7.6 Blinding It will not be possible to blind the investigator to the type of device used. However, 5 minutes after completion of intubation, the operating surgeon (who is blinded to the technique of intubation) will examine the oropharynx and record the bleeding. At the time of intubation, the investigator will record the bleeding as seen on video laryngoscope or fiberscope monitor screen.

7.7 Baseline data Base line data includes gender, age, weight, height, BMI & ASA score Airway assessment includes Mallampati score, thyromental distance, mouth opening, jaw protrusion and neck movement. This is the routine assessment undertaken by anaesthetists as a part of standard preoperative airway assessment.

7.8 Trial assessments

The following data will be collected by one of the investigators:

* Incidence and severity nasal bleeding using nasal trauma score (0= no bleeding, 1=minimal bleeding (only visible traces of blood); 2=moderate bleeding (pooling of blood in the pharynx), 3 = severe bleeding (blood in the pharynx sufficient to impede intubation).
* Nasal intubation smoothness score (0=smooth insertion without any resistance, 1= insertion with slight resistance; 2= insertion with great resistance; and 3= change of nostril for insertion).
* Laryngoscopy time (time from insertion of laryngoscope in the mouth to visualize the vocal cords or from the insertion of fiberscope in the nostril to visulise the vocal cords). In the VL group laryngoscopy is done prior to insertion of tube through the nostril.
* Intubation time (time from insertion of fiberscope or video laryngoscope till first capnography trace)
* Additional manoeuvres required such as tracheal tube impingement, tube rotation, external laryngeal pressure, use of Magill forceps, success rate of nasotracheal intubation.

7.9 Follow-up assessments Patients will be reviewed in the first 3 to 24 hours whilst they are in the hospital as apart standard postoperative visit. No further follow up is required for this study. If any patients report continuing nasal bleed in the postoperative period, a maxillofacial surgeon will be requested to review the patient for further management and any outcome data may be collected up to 72 hours.

7.10 Withdrawal Participants may withdraw from the study at any time without prejudice. Unless a participant explicitly withdraws their consent, data collection will be completed in line with the consent as per this protocol until the end of the study definition. In the rarity of loss of capacity, cancellation of surgery or unforeseen surgical complications; patients data will be collected to the point of withdrawal. If surgery is cancelled, efforts will be made by the research team to re-schedule surgery in a timely fashion to allow continued participation in the study. If this is not feasible, the patient will be withdrawn.

7.11 End of study definition This is defined as the date of completion of the 24 hour post-surgery data collection on which the last patient (patient number 200) is recruited to the study.

8. STATISTICS AND DATA ANALYSIS

8.1 Sample size calculation From a previous study using video laryngoscopes, the incidence of nasal bleeding was 68% We consider flexible fibrescopes will reduce the bleeding by 33% (1/3). For a power of 90% with a significance level of 0.05 we need 186 patients.

8.2 Planned recruitment rate There four theatre lists involving oral procedures take place every week at University Hospital, Coventry. Each list involves 4 to 6 patients and nearly 50% of these patients require nasal intubation. Therefore, it is feasible to recruit nearly 20 patients per month.

8.3 Summary of baseline data and flow of patients The normally distributed base line data such as age, gender, weight and airway assessment parameters between two groups will be compared using students t test. Statical significance is taken as p value <0.05

8.4 Primary outcome analysis Primary outcome measure is nasal trauma score. Student t-test for normally distributed data and a non-parametric test either Mann-Whitney U test or Kruskal- Wallis test would be used, as appropriate for other parameters.

8.5 Secondary outcome analysis Secondary outcome measures include intubation time, nasal intubation smoothness score, laryngoscopy time intubation success rate, sore throat and nasal discomfort. Student t-test for normally distributed data and a non-parametric test either Mann-Whitney U test or Kruskal- Wallis test would be used, as appropriate for other parameters

8.6 Participant population The participant population would include patients scheduled to undergo elective surgery under general anaesthesia. The study intervention duration would be very short, lasting less than five minutes.

8.7 Procedure(s) to account for missing or spurious data As the study duration is short, we are unlikely to lose any patients to follow-up. All care would be taken to record all necessary data during preoperative visit and during intubation. Although rare, the surgical plan may change and/or surgery may be cancelled after recruiting. In total we need 186 patients to detect a significant difference in the nasal trauma score. We have planned to recruit 200 in total to overcome any missing data or loss of follow up.

9. DATA MANAGEMENT 9.1 Data collection tools and source document identification Case Report Forms will be completed at the time of data collection timepoints as the per schedule of events.

9.2 Data handling and record keeping Original Consent forms will be filed into the investigator site file, 1 copy will be provided to participants, and 1 copy will be included in the participants medical notes. Any data collected on the CRF will be stored in the Investigator Site File and then entered at regular interval into the excel sheet on an encrypted NHS computer. The site file is securely kept in the locked filing cabinet in the anaesthetic department office.

9.3 Access to Data Only members of the research team will have access to the raw data set for the duration of the study, direct access will be granted to authorised representatives from the Sponsor, host institution and the regulatory authorities to permit trial-related monitoring, audits and inspections.

9.4 Archiving Following the resolution of queries and confirmation of study close-out by the Chief Investigator, all essential documentation will be transferred to a third-party archiving service, which provides suitable fire and water-resistant facilities. Study files will be archived for a period of 25 years. Access to the study documentation will be restricted to named individuals within the study team with express permission from the Chief Investigator and Sponsor.

10. TRIAL OVERSIGHT 10.1 Role and responsibilities of the Sponsor UHCW has agreed to act as sponsor for this trial and will undertake the responsibilities of sponsor as defined by the UK Policy Framework for Health and Social Care Research and ICH Good Clinical Practice. An authorised representative of the Sponsor has approved the final version of this protocol with respect to the trial design, conduct, data analysis and interpretation and plans for publication and dissemination of results. As sponsor, UHCW provides indemnity for this trial and, as such, will be responsible for claims for any non-negligent harm suffered by anyone as a result of participating in this trial. The indemnity is renewed on an annual basis and will continue for the duration of this study.

10.2 Role and responsibilities of the Funder This trial has received a small grant of £4988 from The Difficult Airway Society, towards the R&D support. The design and management of this trial are entirely independent of the funder.

10.3 Principal Investigator

The Principal Investigator responsibilities include, but are not limited to:

* Ensuring that the study is conducted as set out in the protocol and supporting documents
* Delegating study related responsibilities only to suitably trained and qualified personnel and ensuring that those with delegated responsibilities fully understand and agree to the duties being delegated to them;
* Ensuring that CVs and evidence of appropriate training for all Site staff are available in the Trial Site File
* Ensuring that all delegated duties are captured in the study Delegation Log
* Ensuring all Adverse Events are documented and reported promptly to the Sponsor;
* Accountability for study treatments at their site;
* Ensuring the study is conducted in accordance with ICH GCP principles;
* Allowing access to source data for monitoring, audit and inspection;
* Ensuring that all source data is complete for analysis

  11. MONITORING, AUDIT & INSPECTION The study will be monitored by the Research & Development department at UHCW as representatives of the Sponsor, to ensure that the study is being conducted as per protocol, adhering to Research Governance and GCP. The approach to, and extent of, monitoring will be specified in a trial monitoring plan determined by the risk assessment undertaken prior to the start of the study.

  12. ETHICAL AND REGULATORY CONSIDERATIONS 12.1 Ethical approval and research governance The study will be conducted in compliance the principles of the ICH GCP guidelines and in accordance with all applicable regulatory guidance, including, but not limited to, the UK policy framework for health and social care research. Ethical approval for this study will be sought from the Research Ethics Committee combined with Health Research Authority (HRA) approval. No study activities will commence until favourable ethical opinion and HRA approval has been obtained. A final report at the conclusion of the trial will be submitted to the approving REC within the timelines defined by the committee. Confirmation of capacity and capability will be obtained from the R&D department obtained prior to commencement of the study at all participating sites.

12.2 Peer review The study design was initially discussed in anaesthetic departmental research meeting and approved by the chair of the department. Subsequently, the study abstract was peer reviewed by the UK Difficult Airway Society as part of the grant application. In addition, the study protocol has been further peer reviewed by an external airway expert.

12.3 Public and Patient Involvement The study lay abstract and patient information sheet has been reviewed by the Patients and Public Research Advisory group and the documents been revised as per their guidance.

12.4 Data protection and patient confidentiality The study will comply with the current Data Protection regulations. Participants will be assigned a unique identifier upon enrolment into the study to allow pseudonymisation of patient-identifiable of patient-identifiable data. Access to patient identifiable data will be restricted to members of the study co-ordination team who require it for the performance of their role. Electronic data will be stored on password protected encrypted drives and hard copies of study documents will be stored in locked filing cabinets in secure entry-card protected sites.

12.5 Safety reporting The study is low risk, comparing standard of care interventions and we are not anticipating any adverse events because of study. If any issues occur due to the standard of care interventions, patients will be followed up via standard of care pathway. If any patients develop significant nasal bleeding (nasal trauma score = 3), they will be first reviewed by the maxillofacial surgeon. If necessary, they will be referred to an ENT surgeon for further management. They would then be followed up for a further 72 hours. Any adverse outcomes experienced by patients will be recorded in the CRF and compared in the final analysis.

Any non-compliance or deviations that occur during the study will be reported to Sponsor as per SOP using the appropriate reporting form.

12.6 Dissemination Following completion of study, the results will be presented at departmental QI meeting and presented as abstract at Difficult Airway Society annual scientific meeting. The study will be published at a peer reviewed Anaesthesia journal. A lay person summary will be sent for those participants who expressed their interest to receive the study results.

Appendix 1 Score descriptions for Nasal intubation smoothness score

Nasal Intubation Smoothness Score Nasal Trauma Score

Score Description Score Description 0 Smooth insertion without any resistance 0 No bleeding

1. Insertion with slight resistance 1 Minimal bleeding
2. Insertion with great resistance 2 Moderate bleeding i.e. pooling of blood in the pharynx
3. Necessity to change nostril for insertion after unsuccessful attempt at tube passage on contralateral side 3 Severe bleeding i.e. blood in the pharynx sufficient to impede intubation

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7433945/ Laryngoscopy time: time from insertion of laryngoscope in the mouth to visualise the vocal cords or from insertion of fibrescope in the nostril to visualise the vocal cords.

Intubation time: from insertion of laryngoscope or fibrescope until first capnography trace is obtained. In the VL group, VL must be inserted first and then the tube is inserted via selected nostril.

Nasal discomfort score Score Description nil No nasal discomfort mild Slight nasal discomfort, easily tolerated moderate Nasal discomfort with awareness of symptoms which are bothersome i.e. sneezing, congestion, itching, bleeding severe Active ongoing uncontrolled symptoms on assessment. i e. pain, bleeding https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7433945/

References

1. Abrons RO, Zimmerman MB, El-Hattab YMS. Nasotracheal intubation over a bougie vs. non-bougieintubation: a prospective randomised, controlled trial in older children and adults usingvideolaryngoscopy. Anaesthesia 2017; 72: 1491-500.
2. Morimoto Y, Sugimura M, Hirose Y, Taki K, Niwa H. Nasotra- cheal intubation under curve-tipped suction catheter guidance reduces epistaxis. Canadian Journal of Anesthesia 2006; 53: 295-8
3. Kim YC, Lee SH, Noh GJ, et al. Thermosoftening treatment of the nasotracheal tube before intubation can reduce epistaxis and nasal damage. Anesthesia and Analgesia 2000; 91: 698- 701.
4. El-Seify ZA, Khattab AM, Shaaban AA, Metwalli OS, Hassan HE, Ajjoub LF. Xylometazoline pretreatment reduces nasotra- cheal intubation-related epistaxis in paediatric dental surgery. British Journal of Anaesthesia 2010; 105: 501-5.
5. Bansal T, Singhal S, Dhingra K. A study to evaluate nasotracheal intubation using Airtraq laryngoscope with a bougie and without a bougie. Indian J Anaesth 2022;66:757-62.
6. Collins SR, Blank RS. Fiberoptic intubation: an overview and update. Respir Care. 2014 Jun;59(6):865-78; discussion 878-80. doi: 10.4187/respcare.03012. PMID: 24891196.
7. Hansel, J., Roger, A.M., et al. (2022) Videolaryngoscopy versus direct laryngoscopy for adults undergoing tracheal intubation, Cochrane Database of Systematic Reviews, 4(4), CD011136. Available at https://pubmed.ncbi.nlm.nih.gov/35373840/ (Accessed 5 July 2023)

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 and above, presenting for elective surgical procedures and requiring general anaesthesia and nasal intubation will be invited to take part in the study.

Exclusion Criteria:

* Patients who do not want to take part or do not give consent
* Patients unable to give written consent.
* Patient physical status of ASA 4 and 5,
* Patients deemed to require awake intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Nasal trauma score | 5 minutes
  a score of 0 to 3 will be provided no bleeding, moderate bleeding, or severe bleeding

SECONDARY OUTCOMES:
nasal intubation smoothness score | 2 minutes
  A score of 0 to 3 being given; smooth insertion (0), slight resistance, insertion with great resistance and not possible to insert requiring change of nostril
Total intubation time | 2 minutes
  time in seconds from insertion of fiberscope or video laryngoscope till first capnography trace
Laryngoscopy time | 2 minutes
  time in seconds from insertion of laryngoscope in the mouth to visualize the vocal cords or from insertion of fiberscope in the nostril to visualise the vocal cords
incidence of post operative sore throat | 24 hours
  Number of patients having soret throat in the post operative period
incidence of postoperative nasal discomfort | 24 hours
  number of patients having nasal discomfort in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Cyprian Mendonca, Study Director — University Hopsitals Coventry & Warwickshire NHS Trust

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Background] Collins SR, Blank RS. Fiberoptic intubation: an overview and update. Respir Care. 2014 Jun;59(6):865-78; discussion 878-80. doi: 10.4187/respcare.03012. PMID 24891196
- [Background] Bansal T, Singhal S, Dhingra K. A study to evaluate nasotracheal intubation using Airtraq laryngoscope with a bougie and without a bougie. Indian J Anaesth. 2022 Nov;66(11):757-762. doi: 10.4103/ija.ija_466_22. Epub 2022 Nov 18. PMID 36590192
- [Background] El-Seify ZA, Khattab AM, Shaaban AA, Metwalli OS, Hassan HE, Ajjoub LF. Xylometazoline pretreatment reduces nasotracheal intubation-related epistaxis in paediatric dental surgery. Br J Anaesth. 2010 Oct;105(4):501-5. doi: 10.1093/bja/aeq205. Epub 2010 Aug 3. PMID 20682569
- [Background] Kim YC, Lee SH, Noh GJ, Cho SY, Yeom JH, Shin WJ, Lee DH, Ryu JS, Park YS, Cha KJ, Lee SC. Thermosoftening treatment of the nasotracheal tube before intubation can reduce epistaxis and nasal damage. Anesth Analg. 2000 Sep;91(3):698-701. doi: 10.1097/00000539-200009000-00038. PMID 10960403
- [Background] Morimoto Y, Sugimura M, Hirose Y, Taki K, Niwa H. Nasotracheal intubation under curve-tipped suction catheter guidance reduces epistaxis. Can J Anaesth. 2006 Mar;53(3):295-8. doi: 10.1007/BF03022218. PMID 16527796
- [Background] Abrons RO, Zimmerman MB, El-Hattab YMS. Nasotracheal intubation over a bougie vs. non-bougie intubation: a prospective randomised, controlled trial in older children and adults using videolaryngoscopy. Anaesthesia. 2017 Dec;72(12):1491-1500. doi: 10.1111/anae.14029. Epub 2017 Sep 15. PMID 28921537